CLINICAL TRIAL: NCT04396418
Title: Stroke Prevention and Rhythm Control Therapy: Evaluation of an Educational Programme of the European Society of Cardiology in a Cluster-Randomised Trial in Patients With Atrial Fibrillation
Brief Title: Stroke Prevention and Rhythm Control Therapy STEEER-AF
Acronym: STEEER-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Society of Cardiology (Network)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STEEER-AF
Record Dates: First submitted 2020-05-14; First posted 2020-05-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Guideline adherence; stroke prevention; rhythm control; trial
MeSH Terms: conditions — Atrial Fibrillation | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): A 16-week blended learning programme targeting stroke prevention and rhythm control therapy at the healthcare professional level, with controlled assessments, a commitment to change plan, and reinforcement actions
  Interventions: Behavioral: Education
- Control arm (Other): No added education of healthcare professionals
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Randomization between two groups at site level. One cluster with education and one without.

SUMMARY:
A prospective trial with hospitals/health centres across 6 different European countries, being randomised to either a structured education programme as the intervention or no additional education as the control. To determine whether a comprehensive educational programme for healthcare professionals will increase the rate of appropriate stroke prevention and rhythm control therapy in patients with atrial fibrillation (AF) and adherence to Guidelines.

DETAILED DESCRIPTION:
Prospective, parallel group, two-arm, unblinded, international, cluster-randomized controlled trial.

Intervention arm: A 16-week blended learning programme targeting stroke prevention and rhythm control therapy at the healthcare professional level, with controlled assessments, a commitment to change plan, and reinforcement actions Control arm: No added education of healthcare professionals 70 centres with a cluster size of 25 patients; total estimated number of patients 1750.

8-12 weeks patient recruitment period at each centre; 16 weeks educational intervention period; primary & secondary outcomes at 6-9 months post-randomisation; remote follow-up for clinical events (no new patient contact) at 18 months from randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AF
* Patient consents to data collection at baseline and follow-up.

Exclusion Criteria (patients only):

* Patients aged under 18 years of age,
* Pregnant or planning pregnancy,
* Participating in another clinical trial of an investigational medicinal product or device,
* Life expectancy of less than 2 years.

Patient assessment: Baseline (time of recruitment) and at follow-up routine appointment (6-9 months), plus remote follow-up at 18 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1732 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to ESC Guidelines in Atrial Filbrillation | 25 months per centre
  Full adherence to guidelines for stroke prevention rhythm control therapy

SECONDARY OUTCOMES:
Proportion of relevant guidelines adhered to | 25 months per centre
  Proportion of relevant guidelines adhered to for stroke prevention and rhythm control

OTHER OUTCOMES:
Process outcome | 25 months per centre
  Improvement in knowledge and guideline-adherent practice by healthcare professionals using the educational intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hein Heidbuchel, Study Chair — Universiteit Antwerpen; Dipak Kotecha, Study Director — University of Birmingham; Isabelle van Gelder, Study Director — University Medical Center Groningen, The Netherlands; Serge Boveda, Principal Investigator — Clinique Pasteur, France; Philipp Sommer, Principal Investigator — Ruhr-Universität Bochum, Germany; Giuseppe Boriani, Principal Investigator — University of Modena & Reggio Emilia; Maciej Sterliński, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Luis Mont, Principal Investigator — University of Barcelona, Spain; Kim Rajappan, Principal Investigator — University of Oxford, UK; Eduard Guasch, Principal Investigator — University of Barcelona, Spain
Locations (70):
- France (15):
  - CHU Rennes, Rennes, 'Ille-et-Vilaine, Brittany
  - CHU La Timone, Marseille, Bouches-du-Rhône
  - CHU Dijon - Hôpital du Bocage, Dijon, Burgundy
  - Hôpital Cardiologique du Haut-Lévèque, Pessac, Gironde, Nouvelle-Aquitaine
  - CHU Dupuytren, Limoges, Haute-Vienne
  - CHU Nancy, Hôpitaux de Brabois, Nancy, Meurthe-et-Moselle (Lorraine)
  - CHU Rouen, Rouen, Normandy
  - CHU Rangueil, Toulouse, Occitanie, Haute-Garonne
  - CHU Poitiers, Poitiers, Poitou-Charentes
  - CHU Aix en Provence, Aix-en-Provence, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de Pau, Pau, Pyrénées-Atlantiques
  - CHI Toulon La Seyne-sur-Mer Sainte Musse, Toulon, Var
  - Hôpital Henri Mondor (APHP), Créteil, Île-de-France Region
  - CHU Pitié-Salpetrière, Paris, Île-de-France Region
  - Centre Cardiologique du Nord (CCN), Saint-Denis, Île-de-France Region
- Germany (11):
  - University Hospital Würzburg, Würzburg, Bavaria
  - Segeberger Kliniken GmbH, Bad Segeberg, chleswig-Holstein
  - Herzzentrum Niederrhein Krefeld, Krefeld, North Rhine-Westphalia
  - Heart Centre Bad Neustadt, Neustadt, Rhineland-Palatinate
  - Praxisklinik Herz Und Gefässe, Dresden, Saxony
  - Heart Center Leipzig, University of Leipzig, Leipzig, Saxony
  - Herz Riesa, Riesa, Saxony
  - Asklepios Klinik St. Georg, Hamburg
  - Heart Center University Hamburg, Hamburg
  - Medizinische Hochschule Hannover, MHH, Hanover
  - Universitätsklinikum Schleswig-Holstein Lübeck, Lübeck
- Italy (8):
  - Federico II University Hospital, Naples, Campania
  - S Orsola-Malpighi University Hospital, Bologna, Emilia-Romagna
  - Sant'Anna University Hospital of Ferrara, Ferrara, Emilia-Romagna
  - Policlinico di Modena, University of Modena and Reggio Emilia, Modena, Emilia-Romagna
  - Cardiologia Orvieto, Orvieto, Terni
  - University of Florence & AOU Careggi, Florence, Tuscany
  - Clinica Aritmologica, Universita Politecnica delle Marche, Ancona
  - Cardiology Unit Borgo San Lorenzo and Serristori, Florence
- Poland (12):
  - Toruń Hospital, Torun, Vistula Rive
  - District Chojnice Hospital, Chojnice
  - Scanmed Cardiology Center, Ełk
  - Centrum Opieki Medycznej w Jaroslawiu, Jarosław
  - Polikliniką SPZOZ w Lublinie, Lublin
  - Przasnysz, Przasnysz
  - Pułtusk, Pułtusk
  - Siedlce 2 Hospital, Siedlce
  - Wojewódzki Szpital Specjalistyczny nr 5 im, Sosnowiec
  - Szpital Wojewodzki in Sw. Lukasza / Regional Specialist Hospital, Tarnów
  - Wegrow Hospital, Węgrów
  - Lukow, Łuków
- Spain (11):
  - Hospital Universitario Puerta del Mar, Seville, Andalusia
  - Virgen del Rocio University Hospital, Seville, Andalusia
  - Hospital Miguel Servet, Zaragoza, Aragon
  - Hospital Vall d'Hebron, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, Barcelona, Catalonia
  - Hospital Germans Trias i Pujol, Barcelona, Catalonia
  - Hospital Universitari Doctor Josep Trueta, Girona, Catalonia
  - Hospital General Universitario de Alicante, Alicante, Valencian
  - Hospital Universitario La Paz, Madrid
  - Hospital La Fe.com.Valencianna, Valencia
  - Hospital Gral Vigo, Galicia, Vigo
- United Kingdom (13):
  - Buckinghamshire Healthcare NHS Trust - Wycombe Hospital, Buckingham, Buckinghamshire
  - Norwich Hospital, Norwich, East of England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Homerton Hospital, London, England
  - St Bartholomew's Hospital, London, England
  - Imperial College London Chelsea and Westminster Hospital NHS foundation, London, England
  - James Cook University Hospital, Middlesbrough, England
  - Northampton General Hospital, Northampton, England
  - Royal Berkshire foundation NHS trust, Reading, England
  - York Hospital, York, North Yorkshire
  - Horton General Hospital, Banbury, River Cherwell in Oxfordshire
  - Royal Devon and Exeter NHS Foundation Trust, Exeter, West England
  - Queen Elizabeth II, Birmingham

REFERENCES:
- [Derived] Kotecha D, Bunting KV, Mehta S, Sommer P, Sterlinski M, Rajappan K, Mont L, Guasch E, Boveda S, Boriani G, Sun Y, van Deutekom C, Gale CP, De Potter TJR, van Gelder IC; STEEER-AF investigators. Education of healthcare professionals to improve guideline adherence in atrial fibrillation: the STEEER-AF cluster-randomized clinical trial. Nat Med. 2025 Aug;31(8):2647-2654. doi: 10.1038/s41591-025-03751-2. Epub 2025 Jun 13. PMID 40514462
- [Derived] Sterlinski M, Bunting KV, Boriani G, Boveda S, Guasch E, Mont L, Rajappan K, Sommer P, Mehta S, Sun Y, Gale CP, van Deutekom C, Van Gelder IC, Kotecha D; STEEER-AF Trial Team. Design and deployment of the STEEER-AF trial to evaluate and improve guideline adherence: a cluster-randomized trial by the European Society of Cardiology and European Heart Rhythm Association. Europace. 2024 Jul 2;26(7):euae178. doi: 10.1093/europace/euae178. PMID 38940494
- [Derived] Szymanski P, Weidinger F, Lordereau-Richard I, Himmelmann A, Arca M, Chaves J, Lee C, Jonker C, Kotecha D, O'Kelly J, Plueschke K, Rys A, Segec A, Wallentin L, Veltrop R, James S. Real world evidence: Perspectives from a European Society of Cardiology Cardiovascular Round Table with contribution from the European Medicines Agency. Eur Heart J Qual Care Clin Outcomes. 2023 Feb 28;9(2):109-118. doi: 10.1093/ehjqcco/qcad009. PMID 36746430
- [Derived] Banerjee A, Pasea L, Chung SC, Direk K, Asselbergs FW, Grobbee DE, Kotecha D, Anker SD, Dyszynski T, Tyl B, Denaxas S, Lumbers RT, Hemingway H. A population-based study of 92 clinically recognized risk factors for heart failure: co-occurrence, prognosis and preventive potential. Eur J Heart Fail. 2022 Mar;24(3):466-480. doi: 10.1002/ejhf.2417. Epub 2022 Jan 26. PMID 34969173